CLINICAL TRIAL: NCT01299090
Title: Prospective Pellevé™ Neck Wrinkle Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellman International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEL-09-02
Record Dates: First submitted 2011-02-04; First posted 2011-02-18 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Facial and Neck Rhytides
Keywords: wrinkles; rhytides
MeSH Terms: conditions — Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): All subjects enrolled were in the treatment group.
  Interventions: Device: Pelleve Wrinkle Treatment System - includes the Pelleve Handpiece and S5 generator

INTERVENTIONS:
Device: Pelleve Wrinkle Treatment System - includes the Pelleve Handpiece and S5 generator — two treatments spaced 30 days apart

SUMMARY:
Use of RF device to treat wrinkles of the neck

DETAILED DESCRIPTION:
This is a prospective study evaluating the safety and efficacy of two treatments, spaced at 30 day intervals, using the Surgitron® Dual RF™ S5 with the Pellevé™ wrinkle treatment handpiece and Pellevé™ treatment gel for the treatment of neck wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years of age
* Subjects with clinical evidence of neck wrinkles moderate to severe in severity as specified by a grade 4-9 on the Fitzpatrick Wrinkle Assessment Scale.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Willingness and ability to provide written photo consent and adherence to photography procedures(i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

* Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
* Subjects who have had prior exposure to any hyaluronic acid, or any other filler, injection for any purpose in the 12 months preceding study enrollment through the duration of the study.
* Subjects who have had prior exposure to any botulinum toxin for rhytids in the treatment area in the 6 months preceding study enrollment through the duration of the study.
* Subjects who have had a prior cosmetic procedure to improve rhytids in the treatment area (i.e.,rhytidectomy, CO2/erbium laser resurfacing, Thermage/Thermacool radiofrequency treatment)within 12 months or who have visible scars that may affect evaluation of response and/or quality of photography.
* Microdermabrasion, or prescription level glycolic acid treatments within 3 months prior to study participation or during the study.
* Active cut, wound, or infection on the skin.
* Oral Isotretinon within the past 12 months.
* Active HSV-1.
* History of keloids or hypertrophic scarring.
* Existing or history of skin malignancy in the treatment area during the past 12 months.
* Existing or history of skin disease in the treatment area during the past 12 months.
* History of collagen or vascular disease.
* Subjects who have implantable pacemaker, automatic implantable defibrillator/ cadioversor (AICD), or any other implantable electric device.
* Subjects who have used, within 30 days, any medication that can cause dermal hypersensitivity or affect skin characteristics.
* History of autoimmune disease.
* History of any disease that inhibits pain sensation.
* History of Diabetes I or II.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment or unreliability.
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Chipps, MD, Principal Investigator — Moy-Fincher-Chipps Facial Plastics/Dermatology
Locations (1):
- Moy-Fincher-Chipps Facial Plastics/Dermatology, Beverly Hills, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (8.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Neck and Facial Wrinkles Using the Fitzpatrick Wrinkle Assessment
Description: Three independent investigators blinded to photography time points will perform retrospective evaluations of photography from all visits using the 9-point Fitzpatrick Wrinkle Assessment Scale for assessment of neck and facial wrinkles at the culmination of the study.
  The measurement is for percentage of patients who showed improvement
Time Frame: 90 days post treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 49
percentage of participants | 74

2. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The rate of adverse events will be assessed throughout the duration of the study
Time Frame: 90 days post treatment
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 49
participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No